CLINICAL TRIAL: NCT06656702
Title: Effects of Psilocybin in Patients With Amyotrophic Lateral Sclerosis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00408938
Record Dates: First submitted 2024-10-17; First posted 2024-10-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Other): All subjects will be in the same, open label arm
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin Trihydrate. Participants will complete an 8-week course of study treatment including two psilocybin sessions (15 mg in week 4 and 15 or 25 mg in week 6), with follow-up assessments 1, 3, and 6 months after the final psilocybin session.

SUMMARY:
This study aims to study the feasibility of psilocybin therapy for patients with Amyotropic Lateral Sclerosis (ALS) with depressed mood. The secondary objective is to assess its impact on depression, quality of life, hopelessness, and functional status in this patient population.

DETAILED DESCRIPTION:
The proposed research's primary objective is to study the feasibility of psilocybin therapy for patients with ALS with depressed mood. The secondary objective is to assess its impact on depression, quality of life, hopelessness, and functional status in this patient population. The proposed proof-of-concept interventional trial will use a single-arm design. The study will be an open-label trial in a sample of up to 24 treatment-seeking patients with a diagnosis of ALS and depressed mood. Participants will complete an 8-week course of study treatment including two psilocybin sessions (15 mg in week 4 and 15 or 25 mg in week 6), with follow-up assessments 1, 3, and 6 months after the final psilocybin session.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and older.
2. Patients must fulfill ALS El Escorial criteria for possible, probable, laboratory supported probable or definite ALS.
3. Patients with a pulmonary forced vital capacity (FVC) >60%. The investigators have chosen this measure of function to account for respiratory decompensation during the 6-month longitudinal portion of the study.
4. Patients with ability to swallow tablets by mouth. Participants may have a feeding tube, but must be able to swallow by mouth and cannot use the feeding tube to administer the psilocybin tablet.
5. Clinically significant depressive symptoms as evidenced by an Assessment of Depression Inventory (ADI)-12 score >22.

Exclusion Criteria:

1. Patients with severe speech impairments, including those who are nonverbal, require assisted speech devices, and those who can only communicate by writing or texting.
2. Patients who are unable to consent for themselves.
3. Patients with tracheostomy or continuous continuous positive airway pressure (CPAP) or BiPAP.
4. Known clinical evidence of frontotemporal dementia.
5. Cardiovascular conditions: corrected QT interval (QTc) >450 msec, uncontrolled hypertension (i.e., systolic blood pressure (SBP)> 139 mm Hg, diastolic blood pressure (DBP)> 89 mm Hg), resting heart rate (HR)> 90 beats per minute, angina, a clinically significant ECG abnormality (e.g., atrial fibrillation), transient ischemic attack (TIA) in the last 6 months, stroke, peripheral or pulmonary vascular disease (no active claudication).
6. Epilepsy with history of seizures
7. Renal disease (creatinine clearance <40 ml/min using the Cockraft and Gault equation)
8. Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
9. Females who are pregnant (positive pregnancy test) or nursing, or are not practicing an effective means of birth control (i.e., intrauterine systems/devices, hormonal methods including implant, shot, patch, ring, or oral contraceptive, condom, diaphragm, sterilization, and abstinence).
10. Currently taking medications that interact with psilocybin on a regular (e.g., daily) basis: Atypical antidepressants, such as mirtazapine (Remeron), trazodone (Oleptro), vortioxetine (Brintellix), and vilazodone (Viibryd); Tricyclic antidepressants, such as amitriptyline, imipramine (Tofranil), nortriptyline (Pamelor), desipramine (Norpramin), doxepin, trimipramine (Surmontil), and protriptyline (Vivactil); and Monoamine oxidase inhibitors (MAOIs), such as Selegiline (Emsam), tranylcypromine (Parnate), phenelzine (Nardil) and isocarboxazid (Marplan).
11. Currently taking Nuedexta (dextromethorphan/quinidine combination), efavirenz, Acetaldehyde dehydrogenase inhibitors such as disulfiram (Antabuse), Alcohol dehydrogenase inhibitors, or UGT1A9 inhibitors or UGT1A10 inhibitors such as phenytoin, regorafenib, eltrombopag.
12. Current or history of meeting Diagnostic and Statistical Manual (DSM)-5 criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I Disorder
13. Have a first degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of psilocybin treatment as assessed by number of participants recruited, retained and adhere to treatment | 6 months
  feasibility will be assessed by participant recruitment, retention, and treatment adherence.

SECONDARY OUTCOMES:
Depressive symptoms as assessed by the Montgomery-Asberg Depression Rating Scale | Baseline, 1 week post psilocybin session, 1 month post psilocybin session
  Depressive symptoms from baseline at 1 week and 1 month after final psilocybin session measured by the Montgomery-Asberg Depression Rating Scale. Score range: 0-60; higher scores = worse outcome
Depressive symptoms as assessed by the and ALS Depression Inventory | Baseline, 1 week post psilocybin session, 1 month post psilocybin session
  Depressive symptoms from baseline at 1 week and 1 month after final psilocybin session measured by the ALS Depression Inventory. Score ranges from 12 (best) to 48 (worst), with scores between 23 and 29 indicating mild depression and scores above 30 indicating severe depression.
Impact of psilocybin treatment on quality of life as assessed by the EuroQoL 5-dimension, 3-level (EQ-5D-3L) 5-item ALS Assessment Questionnaire | 6 months
  Impact on quality of life measured by the 5-dimension, 3-level EuroQol, 5-item ALS Assessment Questionnaire. Score range 5-25; higher score more problems. The EQ-5D-3L also includes an EQ VAS, which is a vertical scale where respondents rate their health from "the best health you can imagine" to "the worst health you can imagine". The EQ-5D-3L index is calculated by subtracting the descriptive system values from 1, with 1 representing the best possible health status and a value below 0 representing the worst.
Impact of psilocybin treatment on hopelessness as assessed by the Beck Hopelessness Scale | 6 months
  Impact on hopelessness measured by the Beck Hopelessness Scale. Scores range from 0-20 with higher scores indicating a greater degree of hopelessness.
Impact of psilocybin treatment on function as assessed by the ALS Functional Rating Scale-Revised | 6 months
  Impact of function measured by the ALS Functional Rating Scale-Revised. Scale from 0 = can't do, to 4 = normal ability, with a total score range of 0- 52 points. Higher score better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ambereen K Mehta, MD, MPH, FAAHPM, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Psychedelic and Consciousness Research, Baltimore, Maryland, United States